CLINICAL TRIAL: NCT04005014
Title: Effect of Using Myopia Prediction Algorithm on Children's Eye Refraction in China: a Multi-center Randomized Control Trial
Brief Title: Effect of Using Myopia Prediction Algorithm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CCPMOH2019-China-1
Record Dates: First submitted 2019-07-01; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Eye--Refractive Errors

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Examinations of visual acuity, eye refraction and biometrics will be performed in each participating clinic by trained investigators. The investigators, outcomes assessors involved in data management and analysis will be blinded to the group assignment. The study participants, the coordinator, senior consultants, and study personnel responsible for randomisation will not be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using myopia prediction algorithm (Experimental): After examination of visual acuity, eye refraction and biometrics, the examination results are shown to the children. Meanwhile, myopia prediction algorithm will be used to predict SE and presence of high myopia in the subsequent 10 years.
  Interventions: Other: Myopia prediction algorithm
- Not using myopia prediction algorithm (No Intervention): After examination of visual acuity, eye refraction and biometrics, the examination results are shown to the children.

INTERVENTIONS:
Other: Myopia prediction algorithm — Candidate predictors included age at examination, SE, and annual progression rate. Using these predictors, the algorithm will be used to predict SE and whether patients will progress to high myopia in the subsequent 10 years.
  Arms: Using myopia prediction algorithm

SUMMARY:
In this study, the investigators aim to perform a prospective, randomized controlled study to compare the myopia development between children using myopia prediction algorithm and children without using myopia prediction algorithm.

DETAILED DESCRIPTION:
We propose to enroll Grade 3 children from primary schools in China. Children will be given examinations of visual acuity, eye refraction and biometrics, and be assigned to two groups: participants in group A use myopia prediction algorithm to predict myopia development, while in Group B, the participants do not use myopia prediction algorithm to predict myopia development. The visual acuity, eye refraction and biometrics will be investigated over the one-year follow-up period, aiming at comparison of actual myopia development between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Children at Grade 3 (aged 8-9)
* Has the record of eye refraction examined in the past year
* Written informed consents provided

Exclusion Criteria:

* Definitive diagnosis of other ocular abnormalities except for refractive error
* Previous eye surgery
* Unwilling to participate in this trial

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1680 (Estimated)
Dates: Start 2019-07-08 (Estimated); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of SER development of at least -0.5 dioptres (D) | Up to 1 year
  SER: sphere + ½ 360 cylinder; SER development of at least -0.5 dioptres: SER2 - SER1≤-0.5D; SER1: SER at baseline; SER2: SER up to 1 year

SECONDARY OUTCOMES:
Changes in SER \and AL | Up to 1 year
  Changes in SER \and AL will be calculated; AL: axial length
Changes in proportion of children using atropine | Up to 1 year
  Changes in proportion of children using atropine will be calculated
Changes in proportion of children using orthokeratology lenses | Up to 1 year
  Changes in proportion of children using orthokeratology lenses will be calculated
Changes in proportion of children using spectacles | Up to 1 year
  Changes in proportion of children using spectacles will be calculated
Changes in child's average outdoor activity time per day | Up to 1 year
  Changes in child's average outdoor activity time per day will be calculated
Changes in child's average screen time per day | Up to 1 year
  Changes in child's average screen time per day will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University